CLINICAL TRIAL: NCT05468268
Title: Leveraging the Neural Circuits of Hyper-Memory to Ameliorate Memory Dysfunction in Prodromal Alzheimer's Disease (pAD) - Noninvasive Brain Stimulation for pAD (pADmemory)
Brief Title: Noninvasive Brain Stimulation for pAD
Acronym: pADmemory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi di Trento (Other)
Collaborators: University of Roma La Sapienza (Other); I.R.C.C.S. Fondazione Santa Lucia (Other); University Of Perugia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: UStudidiTrento 2021-004
Record Dates: First submitted 2022-07-01; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer's Disease - MCI
Keywords: Transcranial Magnetic Stimulation; Prodromal Alzheimer's Disease; Memory; TMS-EEG; Electroencephalography

STUDY DESIGN:
Intervention Model Description: Factorial Assignment 40 patients with pAD. Patients randomly assigned to 1 of 2 rTMS protocols (20 pAD participants real rTMS and 20 sham rTMS). Patients will be balanced using MoCA and age matching to create homogeneous groups.
  Protocols:
  1. 20 Hz rTMS
  1. Sham rTMS Patients will undergo a clinical, neuropsychological, and neurophysiological evaluation before the start of treatment (baseline, t0), at the end of the rTMS stimulation phase (t1), after 3 (t2) and 6 months (t3) from the end of treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) We will implement a randomized, non-pharmacological study, with a double-blind certified medical device (neither the patient nor the clinician / researcher who will carry out the evaluations will be aware of the group to which the patient has been assigned).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 Hz rTMS (Experimental): rTMS will be applied to the left dorsolateral prefrontal cortex (left DLPFC). The coil will be placed at the EEG 10-20 International System position of the F3 electrode.
  Stimulation parameters will be rTMS delivery of 1600 pulses divided into blocks: 20 Hz for 2 seconds (40 pulses) followed by 28 seconds of pause, with a stimulation intensity equal to 100% of the motor threshold value at rest.
  Interventions: Device: 20 Hz rTMS
- Sham rTMS (Sham Comparator): Sham rTMS will be administered by applying a 30mm thick piece of wood or plastic to a real TMS coil during "stimulation", and this additional element will be constructed in such a way that it appears to be an integral part of the apparatus such that the patient remains unaware that they are not receiving stimulation. This 30 mm distance is adequate to ensure that the magnetic pulse does not reach the cortex.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: 20 Hz rTMS — rTMS stimulation
  Arms: 20 Hz rTMS
Device: Sham rTMS — Sham stimulation
  Arms: Sham rTMS

SUMMARY:
Episodic memory refers to the conscious recalling of a personal experience and includes information of an event and the context in which the event took place.

This function is the first to be impaired in Alzheimer's disease, a degenerative condition in which pathological changes are found initially in the medial temporal cortex and then spread in the rest of the cortex starting from post-Rolandic areas.

This study aims at examining the mechanisms that enhance memory processes, based on the information acquired by studying hypermnesic subjects. The recent discovery of subjects with an extraordinary ability to remember past events (highly above-average autobiographical memory) and the development of techniques to manipulate memory circuits in rodents provide a unique opportunity to study the mechanisms that determine the facilitation of memories.

As part of a multicenter project funded by the Ministry of Health in collaboration with La Sapienza University of Rome, the University of Perugia and the Santa Lucia Rehabilitation Center in Rome, the aspect of the project carried out at CIMeC (University of Trento) will consist in evaluating the changes induced by rTMS in patients with prodromal Alzheimer's disease, after stimulation of the regions that appear particularly active in hypermnesic subjects.

This project would offer the possibility of accessing an innovative non-invasive, and non-pharmacological treatment.

The specific objectives are:

(i) To evaluate the effectiveness of rTMS applied to hyperactive areas in hypermnesic subjects in enhancing autobiographical memories; (ii) Analyzing the neural correlates of the behavioral variations. The study will allow us to define whether it is possible to improve the recollection of autobiographical events by stimulating the circuits that are more active in hypermnesic subjects.

The results will be crucial to gain a better understanding of the mechanisms through which brain stimulation contributes to the promotion of neuroplasticity and the effects of rTMS in the prodromal stages of Alzheimer's dementia.

DETAILED DESCRIPTION:
METHODS AND PROCEDURES:

Materials and methods of the investigation will be the following:

* repetitive Transcranial Magnetic Stimulation (rTMS)
* A general neuropsychological assessment battery
* Questionnaires and scales
* Electroencephalogram (EEG) recording
* Combined EEG recording and single-pulse TMS (TMS- EEG)

Different rTMS stimulation protocols will be applied:

1. rTMS: this protocol consists in the administration of 1600 pulses at 20 Hz, alternating 2 s of stimulation and 28 seconds of pause. rTMS will be applied over the left dorsolateral prefrontal cortex (left DLPFC). The coil will be placed at the EEG 10-20 International System position of the F3 electrode. The stimulation intensity will be equal to 100% of the motor threshold value at rest. rTMS will be delivered through a Medtronic-Magpro magnetic stimulator and a 70-mm figure-of-eight coil.
2. sham rTMS: as for the protocol that involves the application of sham/placebo stimulation, the rTMS will be administered by applying to the coil a piece of wood or plastic of about 30 mm in thickness, a distance that ensures that the magnetic pulse does not reach the cortex and built so to appear as an integral part of the apparatus.

All stimulation parameters are in accordance with the safety guidelines for the application of rTMS.

Neuropsychological and psychological evaluation:

All patients will undergo a neuropsychological assessment before starting the treatment (baseline=t0=week 1), at the end of the rTMS phase (t1=Week 4), after 3 months (t2=Week 16), and after 6 months (t3=Week 28) from the beginning.

The follow-up evaluation after the end of the treatment will allow verifying long-term effects.

A possible "practice effect" resulting from the frequent and close administration of neuropsychological tests is expected and will be considered in the data analysis, as in all experimental protocols of this type. The practice effect is a common factor for all experimental groups and does not affect the evaluation of the treatment effectiveness.

TMS-EEG data recording: the EEG will be acquired from 64 sintered Ag / AgCl electrodes placed on the scalp in accordance with the international 10-20 system through an EEG acquisition system compatible with TMS. The EEG signal will be acquired with a high-pass filter at 0.01 Hz, a low-pass filter at 1000 Hz, and a sampling frequency of 5000 Hz. The impedance of the electrodes will be kept below 5 kΩ.

The TMS-EEG co-registration will consist of the administration of 180 pulses on the target area stimulated in the application phase of the protocol (left DLPFC), with a random inter-stimulus interval of 2-3 s. rTMS single pulse will be delivered through a Magstim Rapid2 magnetic stimulator (Magstim, Whitland, UK) and a 70-mm figure-of-eight coil.

In the first session, the stimulation hot spot, coil orientation, and TMS intensity will be decided using the rt-TEP software. Specifically, individual stimulation sites (over left DLPFC) will be determined based on the assessed amplitude, morphology, and topography of the average EEG response, following the software developer indications (based on 20-trial average EEG responses to TMS, the investigators will look for a peak-to-peak amplitude near Vpp > 10 µV, in the early 10-50 ms components in the EEG channels located underneath the TMS coil, avoiding the muscle artifacts as much as possible by rotating the coil). During all TMS-EEG recordings, a masking sound, based on the TMS Adaptable Auditory Control -TAAC, will be played via earphones in order to avoid auditory EEG responses evoked by the TMS coil discharge.

The analysis of the data recorded by the combined TMS-EEG will allow an in-depth evaluation of the modulation of cortical activity induced by the different stimulation protocols (real or sham rTMS) and, in particular, will allow investigating cortical excitability and inhibition, connectivity cortico-cortical and the intrinsic ability of the stimulated areas to generate oscillatory activity. This method will provide a unique measure of local cortical activity and effective cortical-cortical connectivity.

STATISTICAL ANALYSIS:

The variables that will be considered for the analysis of neuropsychological and neurophysiological data are:

1. rTMS stimulation effect over time [Prior to treatment (baseline=t0=week 1), at the end of the rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16)]
2. type of stimulation protocol (real or sham rTMS); The experimental design will be both "within-subjects" within each variable of interest (for example, investigating the difference between t1 and baseline to evaluate the effect of rTMS stimulation), and "between subjects" regarding the data between the two stimulation protocols (for example, investigating the difference between real and sham rTMS stimulation).

Correlation analyzes will be performed to identify which neuroplastic changes are linked to improved behavioral performance.

Calculation of sample size:

The primary outcome for the calculation of the sample size was defined as the effect of the rTMS protocol compared to rTMS placebo, on the score achieved at the end of the treatment.

Considering an alpha value of 0.5 - 0,8 and a power of 80% - 95%, the investigators estimate that the number of patients to be recruited should be 14 - 16 patients per group, increased to 20 per group to take into account a possible dropout rate of 20% (pAD participants real stimulation vs. sham stimulation).

Techniques provided for data processing: behavioral and neurophysiological data will be analyzed by analysis of variance (ANOVA) and posthoc comparisons (t-test, contrast analysis).

Statistical processing software: Data processing will be performed using Matlab R2020b (The MathWorks, Massachusetts, USA) and in-house scripts based on functions of the open-source toolbox EEGLAB (https://sccn.ucsd.edu/eeglab/), SPSS and/or Statistica software.

Ethical Considerations and Assessment of the Risk/Benefit Ratio:

Expected benefits: Based on the assumptions of the present project, participants who will receive real rTMS should show a clinical response, based on the primary endpoints reported above, superior to the participants assigned to the sham rTMS protocol. The study also should provide indirect scientific/cognitive benefits, in terms of advancing knowledge on the development of treatments with proven efficacy and on the mechanisms underlying Alzheimer's dementia.

Potential Risks:

The risks are represented by the use of electro-medical devices, that, however, have EC authorization for use with patients. In addition, all the appropriate safety measures will be put in place as indicated by the international scientific community for studies with brain stimulation. Although no adverse events are expected, when the international guidelines for the safe administration of TMS are followed, researchers involved in the project are able to cope with any side effects of stimulation. The stimulation parameters take into account the clinical goals and safety of the participants. Regarding EEG procedures, skin redness immediately under the electrodes is possible, following abrasion from the application of the electroconductive gel.

All the procedures foreseen by the research will be carried out by taking care of the patient, adopting all the necessary measures so that no critical issues related to stress or fatigue arise.

Risk/Benefit Ratio:

In the proposed study, the risk/benefit ratio is in favor of benefit, in terms of increased knowledge and expected direct benefit for the participants.

According to the classification of a consensus paper, this protocol is part of class 2 studies, which identify studies with indirect benefits and moderate risks: these are studies with patients where the clinical benefit is speculative, but from which important data could come for the development of effective treatments.

Ethical Considerations:

At the end of the study, patients will not be informed of the treatment protocol to which they have been assigned but about the overall results of the study, receiving a report containing a summary of the results achieved by the project.

Informed Consent:

Participation in the study is on a voluntary basis: each subject will obtain explicit information regarding the nature of the project and will have to sign a written consent before they can be included. Participants can withdraw their consent to participate at any time, without any consequences and without providing explanation.

Data storage and processing:

The data will be protected and anonymized according to the current procedures. All identification data will be encrypted within the database and the subjects will be identified by a code. However, the nature of the study makes it necessary to maintain the data regarding the identification of the participants because of the follow-up evaluations. Access to the database containing the collected data and the results will be restricted to the researchers involved in the project. Sensitive data and all paper data will be kept under lock and key at CERiN (TMS-EEG laboratory). The research manager will also be responsible for the appropriate conservation of these data. As this study involves experimental data, the experimental data will later be published and shared as aggregated data with national and international scientific communities.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* meet inclusion criteria related to TMS (attached in the protocol)
* to be able to provide information regarding their cognitive and functional skills, or have a caregiver available who is able to provide the patient information necessary for participation in the study and who is present when signing the patient's informed consent.

pAD Patient Inclusion Criteria:

* Clinical Dementia Rating Scale <2;
* Diagnosis of prodromal Alzheimer's disease (amnesic MCI) according to the diagnostic criteria;
* Neurodegeneration biomarker for AD (FDG-PET or CSF), diagnosis confirmed by clinical follow-up;
* Montreal Cognitive Assessment (MoCA) test overall score within the normal limits (equivalent score of 1);
* Absence of severe vascular distress; Patients will be selected through clinical evaluation (battery of neuropsychological tests at the Neurocognitive Rehabilitation Center - CeRiN)

Exclusion Criteria:

* Patients who are unable to perform the tasks required by the experimental procedure;
* History and/or evidence of any other central nervous system disorder that could be interpreted as a cause of dementia such as structural or developmental abnormality, infectious epilepsy, degenerative or inflammatory/demyelinating diseases of the central nervous system such as Parkinson's disease;
* History of significant psychiatric disease which, in the investigator's judgment, could interfere with study participation.
* History of alcohol or other substance abuse, according to DSM-V criteria, if this could be a contributing factor to dementia;
* Presence of cardiac pacemakers, electronic prostheses, bio-stimulators, metal inserts, or electrodes implanted in the brain or skull, or spine;
* Inability to read and /or understand the written information;
* Dermatitis, eczema, extensive scars on the scalp

Absolute exclusion criteria (criteria for TMS)

* presence of cardiac pacemakers, artificial heart valves and/or bio- stimulators;
* presence of hearing aids located in the middle ear;
* presence of metal inserts on the head and shoulders;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
TMS evoked potentials - TEPs changes. Analysis of cortical excitability and inhibition changes | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16)
  180 pulses will be delivered to the target area (left DLPFC) during EEG registration. This outcome will analyze cortical excitability and inhibition changes induced in the state of excitability/inhibition of brain circuits following the TMS impulse. The amplitude will be used as a marker of cortical excitability.
Connectivity Index, cortico-cortical connectivity analysis: changes in the connectivity evoked by TMS | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16)
  180 pulses will be delivered to the target area (left DLPFC) during EEG registration. This outcome will analyze changes in the latencies and topographical distribution of the TEPs thus providing a connectivity index. This connectivity index will be used to infer the propagation of the activity from the stimulation site to functionally connected areas.
TMS evoked oscillations changes | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16)
  180 pulses will be delivered to the target area (left DLPFC) during EEG registration. This outcome will analyze changes in responses induced by TMS in the frequency domain for the intrinsic capacity of the stimulated area to generate oscillatory activity in specific frequency bands
Autobiographical Memory Interview: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  The Autobiographical Memory Interview is a method of assessing autobiographical memory using a text-based analysis of transcribed autobiographical protocols. The script is segmented into internal (temporally and contextually specific) details and external (generic or semantic) details, which are then tallied. Internal scores are conceptualized as reflecting the episodic richness of the mental simulation, whereas external scores include non-episodic components of the mental simulation such as generic information, routine simulations, or verbal artifacts like repetitions.
  Mean changes on test scores: [score ranges min=N/A, max= no limit, higher score=better outcome]
Free and Cued Selective Recall Reminding Test - episodic memory: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Free and Cued Selective Recall Reminding Test: the three measures being evaluated include free recall (the cumulative sum of free recall from the trials; range 0-48), total recall (the cumulative sum of free recall + cued recall from the trials, range 0-48), and cue efficiency (total recall-free recall)/(48-free recall, range 0.0-1.0).
  Mean changes on test scores: [higher score=better outcome]
Montreal Cognitive Assessment Test - cognitive screening: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Scores on the Montreal Cognitive Assessment Test range from zero to 30. A score of 26 and higher is considered normal. If the score is below 25, the result indicates a possible cognitive impairment.
  Mean changes in test scores: [higher score=better outcome]

SECONDARY OUTCOMES:
Raven's Coloured Progressive Matrices™: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of abstract non-verbal reasoning: mean changes in test scores [score range 0-36, higher score=better outcome]
Forward Digit Span and Reverse Digit Span: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of short and long term memory (verbal) - Mean changes in test scores [score range 0-9, higher score=better outcome]
Spatial Span: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of short and long term memory (visuospatial) Mean changes in test scores [score range 0-10, higher score=better outcome]
Prose Memory: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of short and long term memory - Mean changes in test scores [score range 0-28, higher score=better outcome];
Free And Cued Selective Reminding Test: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of short and long-term memory - Mean changes on tests scores [Immediate: score range 0-36; Deferred: score range 0-12, higher score=better outcome]
Rey-Osterrieth Complex Figure and modified Taylor complex figures: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Deferred re-enactment of the Rey-Osterrieth Complex Figure and modified Taylor complex figure: Long-term memory evaluation Mean changes on tests scores [score range 0-36, higher score=better outcome]
Token Test: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the intensive treatment phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t4=Week 28)]
  Evaluation of linguistic production - Mean changes on tests scores [score range 0-36, higher score = better outcome]
Verbal fluency - Semantic fluency and Phonemic fluency: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Mean changes on tests scores: [score range 0-no limits, higher score=better outcome]
Multiple Features Cancellation task: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of attention and executive function (MFCT) - Mean changes in scores on MFCT Time [score range, min= N/A, max= no limit, higher score=worse outcome; Mean changes in scores on MFCT Accuracy [score range min=0, max=20, higher score=better outcome]; Mean changes in scores on MFCT False alarm [score range min: N/A, max= no limit, high score=worse outcome]
Trail Making test (for A, B and B-A conditions): change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of attention and executive function - Mean changes on scores for each condition [score range: min= n/a, max= no limits, higher score=worse outcome]
The Stroop Color and Word Test: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of attention and executive function - Mean changes on scores [score ranges min=N/A, max= no limit, higher score=worse outcome]
Attentional Matrices: change in performance | Prior to treatment (baseline=t0=week 1), at the end of the 10 days rTMS phase (t1=Week 4), 3 months post-treatment (t2=Week 16), & 6 months post treatment (t3=Week 28)]
  Evaluation of attention and executive function - Mean changes on scores [score range 0-60, higher score=better outcome]

CONTACTS AND LOCATIONS:
Overall Officials: Costanza Papagno, MD-PhD, Principal Investigator — Università di Trento, Centro di Riabilitazione Neurocognitiva (CeRiN), Rovereto
Locations (1):
- Centro Interdipartimentale Mente/Cervello (CIMeC); Centro di Riabilitazione Neurocognitiva (CeRiN), Rovereto, Trento, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant's data be available?
  Yes, after deidentification.
  What data will be shared?
  Individual participant's data that underlie the results reported in the article, after deidentification.
  Which other documents will be available?
  The study protocol.
  When will data be available?
  Data will be made available with the article publication, and the period for sharing this data will have no foreseen end date.
  With whom will the data be shared?
  The data will be shared with Investigators whose proposed use of the data has been approved by an independent review committee, for research purposes only.
  For what types of analyses will the data be shared?
  The only data that will be shared will be those that contribute to achieve the research aims of the proposal, previously approved by an independent ethical review committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available with the article publication, and the time frame for sharing this data will have no foreseen end-date.
Access Criteria: Proposals for data sharing should be directed to costanza.papagno@unitn.it following the ethical committee approval. Data requestors need to sign a data access agreement to gain access. The sharing of the data will be contingent on the approval of an independent ethics committee and the relevance of the requested data as it pertains to the research question.

REFERENCES:
- [Background] Bortoletto M, Veniero D, Thut G, Miniussi C. The contribution of TMS-EEG coregistration in the exploration of the human cortical connectome. Neurosci Biobehav Rev. 2015 Feb;49:114-24. doi: 10.1016/j.neubiorev.2014.12.014. Epub 2014 Dec 22. PMID 25541459
- [Background] Casarotto S, Fecchio M, Rosanova M, Varone G, D'Ambrosio S, Sarasso S, Pigorini A, Russo S, Comanducci A, Ilmoniemi RJ, Massimini M. The rt-TEP tool: real-time visualization of TMS-Evoked Potentials to maximize cortical activation and minimize artifacts. J Neurosci Methods. 2022 Mar 15;370:109486. doi: 10.1016/j.jneumeth.2022.109486. Epub 2022 Jan 21. No abstract available. PMID 35074394
- [Background] Chung SW, Rogasch NC, Hoy KE, Fitzgerald PB. Measuring Brain Stimulation Induced Changes in Cortical Properties Using TMS-EEG. Brain Stimul. 2015 Nov-Dec;8(6):1010-20. doi: 10.1016/j.brs.2015.07.029. Epub 2015 Jul 17. PMID 26275346
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Parker ES, Cahill L, McGaugh JL. A case of unusual autobiographical remembering. Neurocase. 2006 Feb;12(1):35-49. doi: 10.1080/13554790500473680. PMID 16517514
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Ferro M, Cincotta M, Ulivelli M, Bartalini S, Miniussi C, Giovannelli F, Passero S. A real electro-magnetic placebo (REMP) device for sham transcranial magnetic stimulation (TMS). Clin Neurophysiol. 2007 Mar;118(3):709-16. doi: 10.1016/j.clinph.2006.11.005. Epub 2006 Dec 22. PMID 17188568
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Kallioniemi, E., Könönen, M., & Määttä, S. (2018). TMS-EEG: Methods and Challenges in the Analysis of Brain Connectivity. Biomedical Engineering Challenges: A Chemical Engineering Insight, 175 https://doi.org/10.1002/9781119296034.ch9
- [Background] Russo S, Sarasso S, Puglisi GE, Dal Palu D, Pigorini A, Casarotto S, D'Ambrosio S, Astolfi A, Massimini M, Rosanova M, Fecchio M. TAAC - TMS Adaptable Auditory Control: A universal tool to mask TMS clicks. J Neurosci Methods. 2022 Mar 15;370:109491. doi: 10.1016/j.jneumeth.2022.109491. Epub 2022 Jan 31. PMID 35101524
- [Background] Sarasso S, D'Ambrosio S, Fecchio M, Casarotto S, Vigano A, Landi C, Mattavelli G, Gosseries O, Quarenghi M, Laureys S, Devalle G, Rosanova M, Massimini M. Local sleep-like cortical reactivity in the awake brain after focal injury. Brain. 2020 Dec 1;143(12):3672-3684. doi: 10.1093/brain/awaa338. PMID 33188680
- [Background] Tulving, E. (1983). Elements of episodic memory.